CLINICAL TRIAL: NCT00724997
Title: Randomized, Double-blind, Placebo-controlled, Phase I Dose-escalation Study of Single Dose GHB01L1 in Healthy Volunteers
Acronym: GHBCS-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVIR Green Hills Biotechnology AG (Industry)
Responsible Party: Thomas Muster PhD, CEO/CSO, AVIR Green Hills Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GHB-CS01; EudraCT 2006-001176-20
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Seasonal Human Influenza
Keywords: live attenuated flu vaccines; Influenza A (H1N1); intranasally application; replication-deficient influenza virus
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- cohort I (Other): dose level I: 6.4 log10 TCID50/volunteer, 8 volunteers randomized at a ratio of 6:2 for GHB01L1 or placebo
  Interventions: Biological: GHB01L1
- cohort II (Other): dose level II: 6.7 log10 TCID50/volunteer, 8 volunteers randomized at a ratio of 6:2 for GHB01L1 or placebo
  Interventions: Biological: GHB01L1
- cohort III (Other): dose level III: 7.0 log10 TCID50/volunteer, 8 volunteers randomized at a ratio of 6:2 for GHB01L1 or placebo
  Interventions: Biological: GHB01L1
- cohort IV (Other): dose level IV: 7.4 log10 TCID50/volunteer, 8 volunteers randomized at a ratio of 6:2 for GHB01L1 or placebo
  Interventions: Biological: GHB01L1
- cohort V (Other): dose level V: 7.7 log10 TCID50/volunteer, 16 volunteers randomized at a ratio of 6:2 for GHB01L1 or placebo
  Interventions: Biological: GHB01L1

INTERVENTIONS:
Biological: GHB01L1 — Study medication administered as a single intranasal aerosol (520ul) at doses of 6.4 log10, 6.7 log10, 7.0 log10, 7.4 log10 and 7.7 log10 TCID50/volunteer
  Other Names: A/New Caledonia/20/99 (H1N1) -like delNS1 virus; GHB01NC(H1N1)

SUMMARY:
The purpose of this phase I trial is to evaluate safety and tolerability of GHB01L1 administered as single dose intranasal aerosol for vaccination against influenza A (H1N1) virus.

This study is performed further to assess local and systemic immune response and to analyse pharmacokinetics (shedding) of a single dose GHB01L1 aerosol administered intranasally.

DETAILED DESCRIPTION:
GHB01L1 intends to provide a novel vaccination for influenza virus infection. Data indicate that the GHB01L1 virus is a promising, safe and immunogenic vaccine candidate with a high protection efficacy against the pathogenic wild-type virus challenge.

48 healthy volunteers will be included in a phase I dose escalation study investigating five dose levels. 8 subjects per each of the five dose levels and additional 8 subjects at the highest dose level respectively the maximum tolerated dose level will be randomized at a ratio of 6:2 for GHB01L1 or placebo according to a fixed dose escalation plan.

After all subjects of one dose level have been treated and observed for the safety observation period of one week, an interim safety review will be performed by an Expert Committee. The Expert Committee will review any occurred adverse event and will decide on dose escalation to the next dose level.

Only male healthy volunteers aged 18-50 and seronegative with respect to the applied virus antigens (with antibody titers <1:10 detected in hemagglutination inhibition assay) will be randomized.

GHB01L1 will be administered once on day 1. After a 3 days inpatient period follow-up visits will be performed on day 4, 5, 8, 15 and the study will be terminated on day 29.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-50 years
* Immune status: seronegative with respect to the applied virus antigens with antibody titres <1:10 detected in the HAI assay with the corresponding antigens)
* Written informed consent to participate in this study

Exclusion Criteria:

* Acute febrile illness (>37.3°C)
* Signs of acute or chronic upper or lower tract respiratory illnesses (sneezing, cough, tonsillitis, otitis etc.)
* History of severe atopy
* Seasonal influenza vaccination 2005/2006, 2006/2007 and/or 2007/2008 and/or pandemic influenza vaccination against H5N1
* Known increased tendency of nose bleeding
* Volunteers with clinically relevant abnormal paranasal anatomy
* Volunteers with clinically relevant abnormal laboratory values
* Simultaneous treatment with immunosuppressive drugs incl. Corticosteroids (≥2 weeks) within 4 weeks prior to study medication application
* Clinically relevant history of renal, hepatic, GI, cardiovascular, haematological, skin, endocrine, neurological or immunological diseases
* History of leukaemia or cancer
* HIV or Hepatitis B or C seropositivity
* Volunteers who underwent rhino or sinus surgery, or surgery of another traumatic injury of the nose within 30 days prior to application of study medication
* Volunteers who have received antiviral drugs, treatment with immunoglobulins or blood transfusions, or an investigational drug within four weeks prior to study medication application
* Volunteers who have received anti-inflammatory drugs 2 days prior to study medication application
* Volunteers who are not likely to cope with the requirements of the study or with a significant physical or mental condition that may interfere with the completion of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of safety and tolerability of GHB01L1 administered as single dose intranasal aerosol will be evaluated by clinical signs and symptoms as well as laboratory tests. | Beginning with signing Informed Consent through 30 days after study end

SECONDARY OUTCOMES:
Local immune response: IgA and cytokines response in nasal mucosal samples. Systemic Immune response: HAI, MNA and IgG assessment in serum samples. Pharmacokinetics: qualitative assessment of viral recovery (shedding) in nasal mucosal samples. | Samples are collected at baseline and at several time points till day 29 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Wacheck, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna General Hospital, Dpmt. of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Morokutti A, Muster T, Ferko B. Intranasal vaccination with a replication-deficient influenza virus induces heterosubtypic neutralising mucosal IgA antibodies in humans. Vaccine. 2014 Apr 7;32(17):1897-900. doi: 10.1016/j.vaccine.2014.02.009. Epub 2014 Feb 22. PMID 24560674
- [Derived] Wacheck V, Egorov A, Groiss F, Pfeiffer A, Fuereder T, Hoeflmayer D, Kundi M, Popow-Kraupp T, Redlberger-Fritz M, Mueller CA, Cinatl J, Michaelis M, Geiler J, Bergmann M, Romanova J, Roethl E, Morokutti A, Wolschek M, Ferko B, Seipelt J, Dick-Gudenus R, Muster T. A novel type of influenza vaccine: safety and immunogenicity of replication-deficient influenza virus created by deletion of the interferon antagonist NS1. J Infect Dis. 2010 Feb 1;201(3):354-62. doi: 10.1086/649428. PMID 20039806